CLINICAL TRIAL: NCT05326048
Title: Defining an Immunological Signature Related to Lesion Location in Multiple Sclerosis
Acronym: APOLLO
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC21_3030_APOLLO
Record Dates: First submitted 2022-03-09; First posted 2022-04-13 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: cytof analysis — cytof analysis of biological samples of CIS patients. Genomic analysis

SUMMARY:
The objective of APOLLO is therefore to identify biomarkers associated with the CNS involvement phenotype in early MS patients.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, retrospective cohort study. In MS patients, a recent study suggests that the location of lesions in the brain relative to the ME is associated with different effector T cell responses (Th17 vs. Th1) to myelin proteins. Thus, lesion localization may be associated with different immune profiles.

Recently, high-resolution techniques such as mass cytometry (CyTOF) have allowed to better decipher immune diversity and thus to identify new potential therapeutic targets. The combination of CyTOF and high dimensional analysis techniques (viSNE, SPADE, MEM) offers robust and reliable methods to identify new subgroups within heterogeneous cell populations. Several studies have explored immune subpopulations by these methods, including B, T, NK or myeloid populations, from peripheral blood or tissues in other pathologies.

Genetic analysis of regions of interest in MS patients could thus allow the establishment of stratification elements potentiating the contribution of immunological markers.

The main objective is to evaluate the relevance of an immunological stratification by CyTOF, allowing the identification of new immune subpopulations associated with the lesion phenotype (brain or brain + ME), in a cohort of MS patients at the beginning of the disease (CIS+) The second objective will focus on genomic profiling of our two groups of MS patients (brain/brain + ME) for different genetic burdens of MS

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically isolated syndrome (CIS) participating in the OFSEP cohort (French MS Observatory)
* At least 18 years old
* Diagnosed with MS according to the 2017 criteria at the time of their last visit
* Not opposed to participating in the study
* Had at least one visit in the year following sampling
* Followed up for at least 1 year after collection.
* Signed OFSEP consent form

Exclusion Criteria:

* CIS patients with progressive MS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CIS patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
Differences in Immune profile | 1 day
  Comparison of immune profile by CyTOF between two groups of MS patients: "brain" versus "brain + ME" CITRUS algorithm will be used to perform a unsupervised hierarchical clustering of cells processed by cytof and SAM test to assess statistical differences in abundances or marker expression levels between groups of patients

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No